CLINICAL TRIAL: NCT02449629
Title: Assessing the Engagement of Transgender and Other Gender Minority Youth Across the HIV Continuum of Care
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 130
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: Transgender, HIV Continuum of Care
Keywords: HIV; Transgender; HIV Continuum of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- TGMY in HIV Care: TGMY (16-24 years of age) currently in HIV care at an Adolescent Medicine Trials Unit (AMTU) site or elsewhere.
- TGMY Not in HIV Care: TGMY (16-24 years of age) not currently in care who are living with HIV, not living with HIV, or those who are unaware of their HIV status.
- Health Care and Social Service Providers: Health care and social service providers who work with TGMY at AMTU sites or elsewhere that serve TGMY within the AMTU cities.

SUMMARY:
This study uses a transformative multiphasic mixed-methods research design that incorporates elements of the following designs:

* Sequential: a secondary data analysis was conducted, using data from ATN 039, ATN 086, and ATN 106, to influence the development of the qualitative interview and quantitative survey instruments for primary data collection.
* Convergent parallel: concurrent collection and analysis of both qualitative and quantitative primary data that will be combined to address the study objectives.

DETAILED DESCRIPTION:
The ultimate goal of this study is to assess engagement of TGMY across the HIV Continuum of Care. This will be accomplished through a transformative multiphasic mixed-methods research study that will engage all sites in the ATN network and collect data from both internal and external sources regarding the facilitators and barriers affecting TGMY's engagement across the HIV Continuum of Care. Empirical and theoretical models will be produced that will guide the future development of HIV-related interventions for TGMY (to be published by the study team in peer-reviewed literature). In addition, findings will be translated into more immediate provider-focused recommendations and multi-media resources that provide concrete guidance and tools that can be applied across socio-ecological levels to promote the full inclusion of TGMY in the various stages of the HIV Continuum of Care. The production of multidisciplinary provider-focused materials that will support the delivery of gender affirming and appropriate HIV care to TGMY is in alignment with many contemporary views of translational research and will have an immediate impact on the ability of providers at AMTU sites and elsewhere to provide HIV-related care to TGMY across the full HIV Continuum of Care.

The research design incorporates elements of both a sequential design (secondary data analysis from ATN 039 and ATN 086/106 influenced the development of measures for primary data collection) and a convergent parallel design (concurrent collection and analysis of both qualitative and quantitative primary data that will be combined to address the specific aims. This design is considered a transformative mixed-methods design due to the study's theoretical and conceptual grounding in Bioecological Systems Theory (BST), Gender Affirmation, and Gender Minority Stress, and the focus on advancing the needs of underrepresented and marginalized populations. Mixed methods studies typically involve collecting and analyzing data derived from both quantitative and qualitative data sources in order to gain greater insight into a research problem than would be gained by using only one of the two methods in isolation. By combining methods, the limitations and biases inherent in one single methodology can be lessened by using multiple forms of data collection. The qualitative phase of the study will use a phenomenological investigative approach, which will help to understand the sociocultural behaviors, language, roles, and interactions within a culture-sharing group (i.e., TGMY) and triangulation of the qualitative data with the quantitative data strengthens the validity of the information received by using a combination of data sources.

ELIGIBILITY:
Inclusion Criteria: Youth Currently in HIV Care

To be considered eligible for enrollment, an individual must meet the criteria listed below.

* Received at least one HIV related service (e.g., medical care, social services, case management, etc.) at an AMTU or elsewhere in the six months prior to consent;
* Does not identify solely with sex assigned at birth (may identify as trans, transgender, trans woman, trans man, man, woman, gender nonconforming, genderqueer, or any other gender, so long as their current gender identity and/or expression do not match their sex assigned at birth);
* Self reports to be HIV-infected;
* Self reports to be between the ages of 16-24 years inclusive at time of consent;
* Ability to understand both written and spoken English;
* Willingness to participate in an in-depth face-to-face qualitative interview about gender minority identity and personal experiences seeking services across the HIV Continuum of Care;
* Willingness to participate in a web-based quantitative survey about gender minority identity and personal experiences seeking services across the HIV Continuum of Care; and
* Able to understand and willing to provide signed informed consent as applicable for study participation.

Exclusion Criteria: Youth Currently in HIV Care To be considered eligible for enrollment, an individual must not meet any of the criteria listed below.

* Active psychiatric condition that, in the opinion of the site personnel, would interfere with the ability to give true informed consent and to adhere to the study requirements;
* Visibly distraught or visibly emotionally unstable (e.g., active hallucinations, exhibiting suicidal, homicidal, or violent behavior) condition that, in the opinion of the site personnel, would interfere with the ability to give true informed consent and to adhere to the study requirements;
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with the ability to give true informed consent and to adhere to the study requirements;
* Acute illness that, in the opinion of the site personnel, would interfere with the subject's ability to adhere to the protocol requirements and/or interfere with the protocol objectives; and
* Site IRB requires parental permission and subject is <18 years of age.

Inclusion Criteria: Youth Not Currently in Care To be considered eligible for enrollment, an individual must meet the criteria listed below.

* Did not receive HIV related services (e.g., medical care, social services, case management, etc.) at an AMTU or elsewhere in the six months prior to the time of consent;
* Does not identify solely with sex assigned at birth (may identify as trans, transgender, trans woman, trans man, woman, man, gender nonconforming, genderqueer, or any other gender, so long their current gender identity and/or expression do not match their sex assigned at birth);
* Self reports to be between the ages of 16-24 years inclusive at time of consent;
* Ability to understand both written and spoken English;
* Willingness to participate in an in-depth face-to-face qualitative interview about gender minority identity and personal experiences seeking services across the HIV Continuum of Care;
* Willingness to participate in a web-based quantitative survey about transgender and other gender minority identity and personal experiences seeking services across the HIV Continuum of Care; and
* Willingness to provide signed informed consent for study participation.

Exclusion Criteria: Youth Not Currently in HIV Care To be considered eligible for enrollment, an individual must not meet any of the criteria listed below.

* Active psychiatric condition that in the opinion of the site personnel would interfere with the ability to give true informed consent and to adhere to the study requirements;
* Visibly distraught or visibly emotionally unstable (e.g., active hallucinations, exhibiting suicidal, homicidal, or violent behavior) condition that, in the opinion of the site personnel interferes with the ability to give true informed consent and to adhere to the study requirements;
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with the ability to give true informed consent and to adhere to the study requirements;
* Acute illness that, in the opinion of the site personnel, would interfere with the subject's ability to adhere to the protocol requirements and/or interfere with the protocol objectives; and
* Site IRB requires parental permission and subject is <18 years of age.

Inclusion Criteria: Health Care and Social Service Providers

To be considered eligible for enrollment, an individual must meet the criteria listed below.

* Fits into one of the following categories: (1) medical provider (physician, nurse, nurse practitioner, physician's assistant); (2) mental health professional (psychologist, psychiatrist, clinical social worker, counselor); (3) case manager/care coordinator; (4) HIV test counselor; (5) or health educator/outreach worker;
* Provides services at one of the 14 AMTU or elsewhere within the AMTU cities; and
* Currently works directly with or has formerly worked directly with TGMY.

Exclusion Criteria: Health Care and Social Service Providers

There are no exclusion criteria.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The three population groups are:
  1. TGMY (16-24 years of age) currently in HIV care at an Adolescent Medicine Trials Unit (AMTU) site or elsewhere.
  2. TGMY (16-24 years of age) not currently in care who are living with HIV, not living with HIV, or those who are unaware of their HIV status.
  3. Health care and social service providers who work with TGMY at AMTU sites or elsewhere that serve TGMY within the AMTU cities.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Types of facilitators that influence the full participation of TGMY in the various stages of the HIV Continuum of Care from the perspective of TGMY with HIV in HIV Care | Entry Visit
  Explore, from the perspective of TGMY living with HIV who are in HIV care, what socio-ecological facilitators exist that influence the full participation of TGMY in the various stages of the HIV Continuum of Care: prevention and testing, diagnosis, linkage to care, engagement in care, retention in care, initiation of ART, adherence to ART, and viral suppression.
Types of barriers that influence the full participation of TGMY in the various stages of the HIV Continuum of Care from the perspective of TGMY with HIV in HIV Care | Entry Visit
  Explore, from the perspective of TGMY living with HIV who are in HIV care, what socio-ecological barriers exist that influence the full participation of TGMY in the various stages of the HIV Continuum of Care: prevention and testing, diagnosis, linkage to care, engagement in care, retention in care, initiation of ART, adherence to ART, and viral suppression.
Types of facilitators that influence the full participation of TGMY in the various stages of the HIV Continuum of Care from the perspective of TGMY not in HIV Care | Entry Visit
  Explore, from the perspective of TGMY who are not in HIV care (including those who are living with HIV, not living with HIV, and those who are unaware of their HIV status), what socio-ecological facilitators exist that influence the full participation of TGMY in the various stages of the HIV Continuum of Care: prevention and testing, diagnosis, linkage to care, engagement in care, retention in care, initiation of ART, adherence to ART, and viral suppression.
Types of barriers that influence the full participation of TGMY in the various stages of the HIV Continuum of Care from the perspective of TGMY not in HIV Care | Entry Visit
  Explore, from the perspective of TGMY who are not in HIV care (including those who are living with HIV, not living with HIV, and those who are unaware of their HIV status), what socio-ecological barriers exist that influence the full participation of TGMY in the various stages of the HIV Continuum of Care: prevention and testing, diagnosis, linkage to care, engagement in care, retention in care, initiation of ART, adherence to ART, and viral suppression.
Types of facilitators that influence the full participation of TGMY in the various stages of the HIV Continuum of Care from the perspective of health care and social service providers | Entry Visit
  Explore, from the perspective of health care and social service providers who provide care and supportive services to TGMY, what socio-ecological facilitators exist that influence the full participation of TGMY in the various stages of the HIV Continuum of Care: prevention and testing, diagnosis, linkage to care, engagement in care, retention in care, initiation of ART, adherence to ART and viral suppression.
Types of barriers that influence the full participation of TGMY in the various stages of the HIV Continuum of Care from the perspective of health care and social service providers | Entry Visit
  Explore, from the perspective of health care and social service providers who provide care and supportive services to TGMY, what socio-ecological barriers exist that influence the full participation of TGMY in the various stages of the HIV Continuum of Care: prevention and testing, diagnosis, linkage to care, engagement in care, retention in care, initiation of ART, adherence to ART and viral suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Harper, PhD, Principal Investigator — University of Michigan
Locations (14):
- United States (14):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Colorado - The Children's Hospital of Denver, Aurora, Colorado
  - Children's Hosp National Med Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Fenway Institute, Boston, Massachusetts
  - Wayne State University-Children's Hospital of Michigan, Detroit, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hopsital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Jadwin-Cakmak L, Reisner SL, Hughto JMW, Salomon L, Martinez M, Popoff E, Rivera BA, Harper GW. HIV prevention and HIV care among transgender and gender diverse youth: design and implementation of a multisite mixed-methods study protocol in the U.S. BMC Public Health. 2019 Nov 15;19(1):1531. doi: 10.1186/s12889-019-7605-4. PMID 31730450
- See also: ATN website — http://www.atnonline.org